CLINICAL TRIAL: NCT00370006
Title: A Phase 1 Clinical Trial to Evaluate the Safety of, and Kinetics and Magnitude of the CMV-Specific Immune Response to, Challenge With a Live Attenuated Strain of CMV (Towne) in Healthy, CMV- Seronegative, Adult Subjects Who Previously Received a CMV Immunotherapeutic Trivalent pDNA Vaccine (VCL CT02) Administered Intradermally or Intramuscularly
Brief Title: Phase 1 Trial of CMV Towne Vaccine in Subjects Previously Received VCL CT02 Vaccine ID or IM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Vical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Jacobson VCL CT-02 IDTC
Record Dates: First submitted 2006-08-28; First posted 2006-08-30 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2006-10

CONDITIONS: Cytomegalovirus Infection
Keywords: cytomegalovirus; vaccine; T cell; antibodies
MeSH Terms: conditions — Cytomegalovirus Infections

INTERVENTIONS:
Biological: Towne CMV vaccine

SUMMARY:
Objectives of this trial are to:

1. Evaluate the kinetics and magnitude of the CMV-specific immune response post-Towne challenge (3000 pfu) in healthy CMV-seronegative volunteers who received VCL CT02 administered ID or IM 9 to 15 months previously as measured by: 1) ELISA and/or virus-neutralizing antibody titers for gB; 2) T-cell IFN-g ELISPOT; 3) T-cell proliferation assays (CFSE) for IE1, pp65, and/or gB; and possibly 4) cytokine and phenotypic flow cytometry responses to pp65, IE1, and/or gB.
2. Evaluate the safety safety of Towne challenge in healthy CMV-seronegative adult subjects who have previously been immunized with a trivalent pDNA CMV vaccine (VCL-CT02) administered intramuscularly (IM) or intradermally (ID).

Our hypothesis is that the immune response to Towne vaccine 3000 pfu challenge after VLC-CT02 priming will be greater than that after Towne vaccination alone (concurrent controls will be administered Towne alone in a concurrent, companion trial).

DETAILED DESCRIPTION:
This is a Phase 1, single-center, open-label trial of the live, attenuated Towne CMV vaccine administered as a "challenge" to healthy, CMV-seronegative, adult subjects who previously received the CMV immunotherapeutic trivalent pDNA-based vaccine, VCL-CT02, given by intradermal or intramuscular routes as described in the following table; these subjects have been followed for 32 weeks.

Table 6.1 Subject Distribution Group Formulation Dosing Regimen (day) Dose per Injection(Administered to the deltoid region) Route of Administration Number of Subjects

1. VCL-CT02 0, 28, 56 1.0 mg Intramuscular (IM) 6
2. VCL-CT02 0, 28, 56 100 μg/injection × 2 injections Intradermal (ID) 11 Total 17

Up to 10 subjects from Groups 1 and 2 will be approached for enrollment in the current protocol. If a subject consents and meets all eligibility criteria, the subject will receive Towne (3000 pfu subcutaneously) between 9 and 15 months after the subject's first dose of VCL-CT02. Safety will be monitored and Both antibody to CMV gB and T-cell responses to CMV antigens will be measured at specified intervals for 252 days post Towne challenge.

ELIGIBILITY:
Inclusion Criteria:18 to 45 years of age at the time of initial enrollment in trial CT02-ID; normal lab values at study entry; good general health; CMV IgG antibody test < 4 times last measured value (i.e., at Week 32 after VCL-CT02 administration in CT02-ID was initiated)

-

Exclusion Criteria:CMV seropositive; recent vaccination(s); immunodeficiency; vaccination with investigational CMV vaccine(s) other than VCL-CT02 ; pregnant or breast-feeding

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10
Dates: Start 2006-09; Study Completion 2007-08

PRIMARY OUTCOMES:
CMV-specific immune response post-Towne challenge: gB antibody, T-cell IFN-g ELISPOT, T-cell proliferation assays for IE1, pp65, and/or gB, cytokine and phenotypic flow cytometry responses to pp65, IE1, gB.

SECONDARY OUTCOMES:
Safety of Towne challenge in subjects who have previously been immunized with a trivalent pDNA CMV vaccine (VCL-CT02).

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Jacobson, MD, Principal Investigator — University of California, San Francisco